CLINICAL TRIAL: NCT02015988
Title: Effectiveness and Tolerability of Early Initiation of Combined Lipid -Lowering Therapy Included Simvastatin and Fenofibrate vs Simvastatin Alone in Patients With Type 2 Diabetes Mellitus, Hypertriglyceridemia and Acute Coronary Syndrome
Brief Title: Simvastatin and Fenofibrate vs Simvastatin Alone in Patients With Type 2 Diabetes Mellitus and Acute Coronary Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Koval' O., MD (Other)
Responsible Party: Sponsor-Investigator, Koval' O., MD, PhD, Professor, Dnipropetrovsk State Medical Academy
Organization: Dnipropetrovsk State Medical Academy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A14-284
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus, Type 2; Hypertriglyceridemia
Keywords: Acute coronary syndrome; Diabetes Mellitus, Type 2; Hypertriglyceridemia; Simvastatin; Fenofibrate
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus, Type 2; Hypertriglyceridemia | interventions — Fenofibrate; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin and Fenofibrate (Experimental): Simvastatin 40 mg once daily and fenofibrate 145 mg once daily orally for 52 weeks (1 year)
  Interventions: Drug: Fenofibrate; Drug: Simvastatin
- Simvastatin (Active Comparator): Simvastatin 40 mg once daily orally for 52 weeks (1 year)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Fenofibrate
  Other Names: Tricor
  Arms: Simvastatin and Fenofibrate
Drug: Simvastatin
  Other Names: Zocor-forte

SUMMARY:
To test the hypothesis that early (within 5-21 days after index event) administration of combined lipid-lowering therapy in extremely high risk population of patients with type 2 diabetes mellitus (T2DM) and hypertriglyceridemia (HTG) who experienced acute coronary syndrome (ACS) will be effective and well tolerated in achievement of contemporary strict requirements for triglyceride (TG) levels as an independent risk factor in the case of HTG with diabetes.

DETAILED DESCRIPTION:
The primary objective of this parallel group study is to demonstrate that the combined therapy of simvastatin and fenofibrate is superior compared to monotherapy with simvastatin based on the comparisons of change of TG levels after 12 weeks of treatment compared to baseline.

Secondary objectives are to compare both treatment alternatives the combination therapy of simvastatin and fenofibrate to simvastatin monotherapy with respect to achievement the European Society of Cardiology 2011 (ESC 2011) non-HDL-C target (less than 2,6 mmol/l), change of apolipoprotein B/apolipoprotein A1 (apoB/apoA1) ratio, High-Density Lipoprotein-Cholesterol (HDL-C), Low-Density Lipoprotein-Cholesterol (LDL-C) and Uric Acid (UA) after 12 weeks and 52 weeks (1 year) of treatment compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Fasting triglycerides ≥ 1,7 mmol/l
* Acute coronary syndrome at least before 5 and maximum 21 days before the inclusion
* If previously treated with statin therapy, the dose should be equivalent to 40 mg of simvastatin at inclusion
* In case of previous statin therapy, last LDL-C measurement before event should be ≤ 2,6 mmol/l
* Written informed consent obtained

Exclusion Criteria:

* Heart failure IV class (NYHA)
* Acute decompensated heart failure
* Life expectancy no more than 1 year
* Chronic kidney disease (CKD) with Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m2
* Severe chronic liver diseases with Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) > 3 Upper Limit of Normal (ULN)
* Known gallbladder disease, including cholecystolithiasis
* Creatinphosphokinase (CPK) > 5 ULN at baseline
* Chronic or acute pancreatitis with the exception of acute pancreatitis due to severe hypertriglyceridemia
* Known photoallergy or phototoxic reaction during treatment with fibrates or ketoprofen,
* Known allergy to peanut or arachis oil or soya lecithin or related products
* Hypersensitivity to simvastatin or fenofibrate or to any of the excipients of the investigational drugs
* Concomitant administration of potent cytochrome P450 isoenzyme 3A4 inhibitors (e.g. itraconazole, ketoconazole, fluconazole, posaconazole, Human Immunodeficiency Virus (HIV) protease inhibitors (e.g. nelfinavir), erythromycin, clarithromycin, telithromycin and nefazodone)
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-09 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in triglycerides (TG) at week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Percentage of patients who achieved non-High-Density Lipoprotein-Cholesterol (non-HDL-C) level less than 2,6 mmol/l at week 12 | Week 12
Percentage changes from baseline in apoB/apoA1 ratio at week 12 | Baseline, Week 12
Percentage changes from baseline in non-High-Density Lipoprotein-Cholesterol (non-HDL-C) at week 12 | Baseline, Week 12
Percentage changes from baseline in High-Density Lipoprotein-Cholesterol (HDL-C) at week 12 | Baseline, Week 12
Percentage changes from baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) at week 12 | Baseline, Week 12
Percentage changes from baseline in uric acid at week 12 | Baseline, Week 12
Percentage of patients who achieved non-High-Density Lipoprotein-Cholesterol (non-HDL-C) level less than 2,6 mmol/l at week 52 | Week 52
Percentage changes from baseline in apoB/apoA1 ratio at week 52 | Baseline, Week 52
Percentage changes from baseline in non-High-Density Lipoprotein-Cholesterol (non-HDL-C) at week 52 | Baseline, Week 52
Percentage changes from baseline in High-Density Lipoprotein-Cholesterol (HDL-C) at week 52 | Baseline, Week 52
Percentage changes from baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) at week 52 | Baseline, Week 52
Percentage changes from baseline in uric acid at week 52 | Baseline, Week 52

OTHER OUTCOMES:
Number of adverse events (AE) caused discontinuations of investigational products | Up to 52 week

CONTACTS AND LOCATIONS:
Overall Officials: Olena A Koval', MD, PhD, Principal Investigator — State Institution "Dnipropetrovsk Medical Academy of Health Ministry of Ukraine"
Locations (1):
- State Institution "Dnipropetrovsk Medical Academy of Health Ministry of Ukraine", Dnipropetrovsk, Ukraine